CLINICAL TRIAL: NCT07080528
Title: Measuring of the Duration of Action of Different Doses of Rocuronium-induced Neuromuscular Block in Infants During Surgical Treatment of Craniosynostosis - a Prospective, Case-controlled Study
Brief Title: Measuring of the Duration of Action of Different Doses of Rocuronium-induced Neuromuscular Block in Infants During Surgical Treatment of Craniosynostosis
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Tamas Vegh, MD (Other)
Responsible Party: Sponsor-Investigator, Tamas Vegh, MD, MD PhD assistant professor, Head Division of General, Transplantation, Vascular and Thoracic Anesthesia, University of Debrecen
Organization: University of Debrecen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AITT 2023/8; 2024-515545-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-24; First posted 2025-07-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Neuromuscular Blocking Agents; Residual Neuromuscular Block; Neuromuscular Blockade Monitoring
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of inhaled anaesthetics on muscle relaxants (Experimental): Duration of action of rocuronium bromide under anaesthesia maintained with Sevoflurane
  Interventions: Drug: Sevofluorane
- Effect of intravenous anaesthetics on muscle relaxants (Experimental): Duration of action of rocuronium bromide under anaesthesia maintained with Propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevofluorane — Investigation of the effect of Sevoflurane on muscle relaxation
  Arms: Effect of inhaled anaesthetics on muscle relaxants
Drug: Propofol — Investigation of the effect of Propofol on muscle relaxation
  Arms: Effect of intravenous anaesthetics on muscle relaxants

SUMMARY:
The use of intravenous muscle relaxants during anaesthesia can significantly facilitate endotracheal intubation and reduce the chance of possible airway complications during intubation. Overall, muscle relaxants make anaesthesia safer. Quantitative measurement of neuromuscular block is essential when anaesthesiologists use muscle relaxants. It allows to avoid postoperative residual block complications such as upper airway obstruction, hypoxia, pharyngeal dysfunction, aspiration.

Unfortunately, quantitative monitoring of neuromuscular block is not routinely used in everyday practice - and this is particularly true in the infant and child population. In adults, the relative absence of easy-to-use and reliable monitors has led to the neglect of neuromuscular monitoring. One of the monitoring techniques suitable for this purpose is electromyography. This EMG-based instrument (TetraGraph ® ) measures the action potential of the musculus adductor pollicis or the musculus abductor digiti minimi muscles.

Clinical trials have shown that for quantitative monitoring of the effect of muscle relaxants, extubation is safe if the TOF ratio is 0.9. Some studies have shown that TOF ratio of 0.95 is necessary to reduce the risk of postoperative respiratory complications.

In this study, investigators will use an EMG-based neuromuscular monitor, the TetraGraph ®, and an electrode specially designed for the infant and child population to measure the muscle relaxant (rocuronium) effect of infants undergoing decompressive surgery for craniosynostosis, from the time of induction until the TOF ratio of 0.9 is reached, using inhaled anaesthetic or intravenous agent to maintain anaesthesia.

In adult population it has been clearly demonstrated that inhaled anaesthetics potentiate the effect of muscle relaxants during maintenance anaesthesia, whereas this effect is moderate or negligible when intravenous maintenance agents are used. There is limited literature on the efficacy of rocuronium in the infant population when anaesthesia is maintained with sevoflurane or propofol. The aim of present study is to improve postoperative patient safety in the infant population.

Infants undergoing anaesthesia for elective craniosynostosis surgery are included in the study. The surgical preparation, anaesthesia of the patients, will be carried out in all aspects according to the daily routine, i.e.: All infants will receive 0.1 mg/kg midazolam i.v. for pre-medication. In the operating theatre, a peripheral vein is provided. Precordial ECG, pulse oximetry, blood pressure measurement, end-expiratory CO 2 , end-expiratory oxygen measurement will be performed during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* 20 infants whose parents have given informed written consent to participate in the studies;
* Age: 3-12 months;

Exclusion Criteria:

* diseases affecting neuromuscular function (myopathies, severe liver and kidney failure);
* Lack of parental consent
* Known allergy to any of the products used

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Time till TOF ratio of 0.9 | From administration of rocuronium to achieve TOF ratio 0.9, during a surgical procedure due to craniosynostosis.
  The primary end point will be to compare the time needed to reach TOFR 0.9 after a single, 0.6 mg/kg dose of rocuronium in anaesthesia maintained by propofol and sevoflurane

SECONDARY OUTCOMES:
Time til TOF count 1, 2, 3, 4 | From the administration of rocuronium to achieve TOF count 1, 2, 3, 4, during a surgical procedure due to craniosynostosis.
  Secondary end points will be the reappearance times for T1, T2, T3 and T4 in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Béla Fülesdi, MD PhD Full Professor DSc, Principal Investigator — University of Debrecen, Faculty of Medicine, Department of Anaesthesiology and Intensive Care
Locations (1):
- University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs-Buder T, Tassonyi E. Intubating conditions and time course of rocuronium-induced neuromuscular block in children. Br J Anaesth. 1996 Sep;77(3):335-8. doi: 10.1093/bja/77.3.335. PMID 8949805
- [Background] Blobner M, Hunter JM, Meistelman C, Hoeft A, Hollmann MW, Kirmeier E, Lewald H, Ulm K. Use of a train-of-four ratio of 0.95 versus 0.9 for tracheal extubation: an exploratory analysis of POPULAR data. Br J Anaesth. 2020 Jan;124(1):63-72. doi: 10.1016/j.bja.2019.08.023. Epub 2019 Oct 10. PMID 31607388
- [Background] Fuchs-Buder T, Brull SJ, Fagerlund MJ, Renew JR, Cammu G, Murphy GS, Warle M, Vested M, Fulesdi B, Nemes R, Columb MO, Damian D, Davis PJ, Iwasaki H, Eriksson LI. Good clinical research practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents III: The 2023 Geneva revision. Acta Anaesthesiol Scand. 2023 Sep;67(8):994-1017. doi: 10.1111/aas.14279. Epub 2023 Jun 22. PMID 37345870
- [Background] Nemes R, Lengyel S, Nagy G, Hampton DR, Gray M, Renew JR, Tassonyi E, Fulesdi B, Brull SJ. Ipsilateral and Simultaneous Comparison of Responses from Acceleromyography- and Electromyography-based Neuromuscular Monitors. Anesthesiology. 2021 Oct 1;135(4):597-611. doi: 10.1097/ALN.0000000000003896. PMID 34329371
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Fuchs-Buder T, Romero CS, Lewald H, Lamperti M, Afshari A, Hristovska AM, Schmartz D, Hinkelbein J, Longrois D, Popp M, de Boer HD, Sorbello M, Jankovic R, Kranke P. Peri-operative management of neuromuscular blockade: A guideline from the European Society of Anaesthesiology and Intensive Care. Eur J Anaesthesiol. 2023 Feb 1;40(2):82-94. doi: 10.1097/EJA.0000000000001769. Epub 2022 Nov 15. PMID 36377554
- [Background] Zarour S, Constantini S, Roth J, Friedman S, Kirgner I, Cohen B, Ekstein M. Postoperative coagulopathy among otherwise healthy pediatric patients undergoing open craniosynostosis repair: a retrospective study. Eur J Pediatr. 2023 Mar;182(3):1341-1349. doi: 10.1007/s00431-023-04805-8. Epub 2023 Jan 14. PMID 36639535
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36639535/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36377554/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18635478/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34329371/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37345870/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31607388/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/8949805/
- Available data/document: Study Protocol — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2024-515545-41-00